CLINICAL TRIAL: NCT02675335
Title: Accelerated Wound Healing in Diabetic Ulcers by Sitagliptin
Acronym: SitaDFU
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Wolfgang-Michael Franz (Other)
Responsible Party: Sponsor-Investigator, Wolfgang-Michael Franz, Professor, Medical University Innsbruck
Organization: Medical University Innsbruck (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SitaDFU_v1.0; 2015-005226-19 (EudraCT Number); MISP 52815 (Other: Merck Investigator Studies Program)
Record Dates: First submitted 2016-02-03; First posted 2016-02-05 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Diabetic Foot
Keywords: Diabetic foot ulcer, Sitagliptin
MeSH Terms: conditions — Diabetic Foot | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin (Active Comparator): Sitagliptin tablets, 100mg per day, 12 weeks treatment
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): Placebo tablets, 1 tablet per day, 12 weeks treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin
  Other Names: Chemical Abstracts Service (CAS) number 654671-77-9
  Arms: Sitagliptin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to test the effect of Sitagliptin on the healing of stable, nonhealing diabetic foot ulcers. This is a randomized placebo-controlled Trial.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* at least 1 diabetic foot ulcer with a size between 1 and 20 sqcm
* stable size of the foot ulcer for at least 2 weeks
* HbA1c <= 8% under Treatment with Insulin, metformin, sulfonylureas, SGLT2 Inhibitors, glinides or glitazones

Exclusion Criteria:

* local purulent signs of Inflammation at ulcer site
* planned interventional or surgical therapy of a macro vessel disease of the lower limb
* glomerular filtration rate <30ml/min
* liver cirrhosis CHILD B or C
* pregnancy, lactation
* allergy against Sitagliptin
* ongoing treatment with dipeptidyl peptidase 4 (DPP4) Inhibitors

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
mean ulcer size after a treatment period of 12 weeks | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang-M Franz, M.D., Principal Investigator — Medical University of Innsbruck

IPD SHARING:
Plan to Share IPD: No